CLINICAL TRIAL: NCT01812733
Title: An Observational Study of Quality of Life, Resource Use and Costs Associated With Treatment of Severe Pain - a Comparison of a Combination of Oxycodone and Naloxone (Targiniq) Versus Oxycodone and Laxatives
Brief Title: Non-interventional Study Comparing Targiniq and Oxycodone/Laxatives
Status: Completed | Type: Observational
Sponsor: Mundipharma AB (Industry)
Responsible Party: Sponsor
Other Study IDs: OXN9513
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Pain; Opioid Induced Constipation
MeSH Terms: conditions — Pain; Opioid-Induced Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the non-interventional study is to compare the quality of life, health care resource use and costs between the use of a combination of oxycodone and naloxone (Targiniq) versus oxycodone and laxatives for patients with severe pain, and to evaluate the cost-effectiveness of treatment with Targiniq.

ELIGIBILITY:
Inclusion criteria:

* Male or non-pregnant female ≥18 years of age
* Malignant or non-malignant opioid sensitive pain
* Must sign an informed consent form (ICF)
* Must have a stable daily dose of oxycodone prolonged release formulation titrated to analgesic effect (as to be assessed by clinical experts)
* Use of laxatives for concomitant opioid-induced constipation in an adequate dose and length of time and without sufficient effect
* BFI ≥30 and state a discomfort caused by the constipation at screening
* Ability to answer the patient questionnaires and have an estimated overall life expectancy of at least six (6) months

Exclusion criteria:

* History of, or on-going, abuse of alcohol and/or drugs
* Inability to read and understand written instructions, ICF or questionnaires
* Constipation not related to opioid use
* Unsuitable patient for other reason(s) in the opinion of the investigator
* Inpatients, if admission and/or discharge is expected during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients have severe pain treated with opioids and will be enrolled at different clinics in Sweden
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 8 Weeks
  Two visits performed over 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabiliteringsmedicinska kliniken, Örebro, Sweden